CLINICAL TRIAL: NCT04452019
Title: Responses on Use of Standing Frame and "Innowalk Pro" in Subacute Patients With Severe Functional Deficits Due to Acquired Brain Injury.
Brief Title: Use of Standing Frame and "Innowalk Pro" in Patients With TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnaas Rehabilitation Hospital (Other)
Collaborators: Made for Movement (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REK106287
Record Dates: First submitted 2020-04-28; First posted 2020-06-30 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2022-11

CONDITIONS: Brain Injuries
Keywords: standing; blood pressure; heart rate; surface electromyography of muscles in legs; perceived exertion
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: All together each included patient will attend five sessions. First session includes an orthostatic test and other baseline measurements. In order to describe test-to-test variation (reliability) when using the devices, two sessions are held in standard standing frame (A) and two sessions in "Innowalk Pro" (B), preferably within the same week. If, for practical reasons, this is not feasible, training is allowed in the following week. The order of the workouts is block randomized to ABAB or BABA at inclusion. The orthostic test and the training session are estimated to last approx. 1 hour including all measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standing frame (Active Comparator): Use of standard standing frame
  Interventions: Device: Use of standard standing frame; Device: Use of a new device; Innowalk Pro
- "Innowalk Pro" (Experimental): Use of a new device; "Innowalk Pro"
  Interventions: Device: Use of standard standing frame; Device: Use of a new device; Innowalk Pro

INTERVENTIONS:
Device: Use of standard standing frame — Two training sessions in a standard standing frame, max 30 min. pr. session
Device: Use of a new device; Innowalk Pro — Two training sessions in Innowalk Pro, max 30 min pr. session

SUMMARY:
This study will explore physical and physiological responses to mobilization of patients with acquired brain injuries in subacute phase using a classic standing frame and a standing device with simultaneous passive movement of legs, "Innowalk Pro".

DETAILED DESCRIPTION:
Several studies underline the importance of early mobilization of patients with brain injuries, leading to shorter hospital stays, less contractures, and improved general function.

The routine mobilization treatment in the rehabilitation of patients with severe brain injuries in Sunnaas Rehabilitation Hospital is initial use of a tilt table where tilt angle is gradually increased, and when tolerated, standing in a classic standing frame where the patient's lower body is fixed to the device in an upright standing position.

"Innowalk Pro" is a robotic standing device where legs are fixed, but passively moved by electric motors in an upright standing position. An assumption is that standing in "Innowalk Pro" might be better tolerated at an earlier stage of rehabilitation than standing in a classic standing frame.

ELIGIBILITY:
Inclusion Criteria:

* Severe brain injury / stroke <1 year post injury.
* Medically stable
* Paresis in lower extremities, minimal walking function (even with personal assistance) (FIM movement (walk), score 1-2)
* Planned stay in Sunnaas RH for a minimum of 2 weeks from time of inclusion
* Tolerate 5 minutes in 40 degrees 'upright' position in tilt table (custom orthostasis test)
* Body weight ≤95 kg
* Body height ≤190 cm

Exclusion Criteria:

* Fractures in the lower extremities or in the columna with movement or strain restrictions or with pain.
* Aggressive and provocative behavior that affects the ability to collaborate.
* Other conditions where upright position is contraindicated

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Standing time in minutes | Up to one week
  Tolerated maximal standing time in each standing device.
Blood pressure | Up to one week
  Blood pressure is monitored continuously

SECONDARY OUTCOMES:
Heart rate | up to one week
  Heart rate will be monitored continuously 5 minutes before and during intervention with Polar 5000
Muscle activity in legs | up to one week
  Any muscle activity in legs during standing session will be monitored by EMG using "Musclelab" (from "Ergotest Innovations") on vastus medialis, hamstrings, tibialis ant. and gastrocnemius muscles.
Spasticity | up to one week
  Spasticity in knee flexors and ankle flexors will be measured by Modified Ashworth scale (0-4 where 0= no increase in tone and 4 = rigid limb)
Perceived exertion | up to one week
  For patients who are cognitive capable, perceived exertion will be registrated on Borg Scale of perceived exertion
Number of patients reporting pain | up to one week
  Negative impact during training
Rate of skin issues | up to one week
  The number of patients reporting
Number of near faints will be registered by the staff. | up to one week
  Negative impact during training

CONTACTS AND LOCATIONS:
Overall Officials: Vivien Jørgensen, Phd, Principal Investigator — Sunnaas Rehabilitaion Hospital
Locations (1):
- Sunnaas Rehabilitation Hospital, Nesoddtangen, Norway

IPD SHARING:
Plan to Share IPD: Yes
Anonymous IPD will be available on request.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available when study has been competed.
Access Criteria: Requests will be reviewed by the Project group.

REFERENCES:
- [Background] Glickman LB, Geigle PR, Paleg GS. A systematic review of supported standing programs. J Pediatr Rehabil Med. 2010;3(3):197-213. doi: 10.3233/PRM-2010-0129. PMID 21791851
- [Background] Riberholt CG, Lindschou J, Gluud C, Mehlsen J, Moller K. Early mobilisation by head-up tilt with stepping versus standard care after severe traumatic brain injury - Protocol for a randomised clinical feasibility trial. Trials. 2018 Nov 8;19(1):612. doi: 10.1186/s13063-018-3004-x. PMID 30409170
- [Background] Riberholt CG, Thorlund JB, Mehlsen J, Nordenbo AM. Patients with severe acquired brain injury show increased arousal in tilt-table training. Dan Med J. 2013 Dec;60(12):A4739. PMID 24355448
- [Background] Frazzitta G, Zivi I, Valsecchi R, Bonini S, Maffia S, Molatore K, Sebastianelli L, Zarucchi A, Matteri D, Ercoli G, Maestri R, Saltuari L. Effectiveness of a Very Early Stepping Verticalization Protocol in Severe Acquired Brain Injured Patients: A Randomized Pilot Study in ICU. PLoS One. 2016 Jul 22;11(7):e0158030. doi: 10.1371/journal.pone.0158030. eCollection 2016. PMID 27447483
- [Background] Piene Wesche A, Strand LI, Jorgensen V, Opheim A, Hoyer E. Early mobilization of a patient with acquired brain injury using a new standing aid, the Innowalk Pro. A single subject experimental design. Disabil Rehabil Assist Technol. 2023 May;18(4):407-414. doi: 10.1080/17483107.2020.1860143. Epub 2020 Dec 23. PMID 33355016
- See also: WESCHE, A.P 2015 Master thesis in Norwegian. "Tidlig mobilisering av voksne pasienter med ervervet hjerneskade ved bruk av "Innowalk Pro". — http://bora.uib.no/handle/1956/11981
- See also: "Innowalk Pro" — https://www.madeformovement.com/innowalk-pro